CLINICAL TRIAL: NCT03420755
Title: Integrating Text Messages Into the Mothers and Babies Course to Address Depression in Low-Income Women and Their Partners
Brief Title: Integrating Text Messages Into the Mothers and Babies Course
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Darius Tandon, Associate Professor, Northwestern University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: STU00203918-A; 1R21MD011320-01 (NIH)
Record Dates: First submitted 2018-01-29; First posted 2018-02-05 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Perinatal Depression; Postpartum Depression
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Intervention Model Description: The investigators will use a stepped wedge design-a form of RCT that involves sequential, but random, rollout of the intervention over multiple time periods. The investigaotrs have created two HV program clusters. Both clusters will initially implement MB 1-on-1 and will recruit MB participants for one quarter (i.e., three months) before crossing over to recruit MB-TXT participants for one quarter. MB-TXT's core curriculum is identical to MB 1-on-1 and adds a series of text messages throughout the curriculum.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MB 1-on-1 Only (Experimental): Mothers and Babies 1-on-1. MB 1-on-1 -12-session intervention Each MB session lasts 15-20 minutes and is delivered as part of a regularly scheduled home visit (English or Spanish).
  Interventions: Behavioral: Mothers and Babies 1-on-1
- MB 1-on-1 Plus TEXT (Experimental): Mothers and Babies Plus Text. MB 1-on-1 along with text enhancements both in English and Spanish.
  Interventions: Behavioral: Mothers and Babies Plus Text

INTERVENTIONS:
Behavioral: Mothers and Babies 1-on-1 — MB 1-on-1 is a 12-session intervention divided into five modules. An introductory 2-session module establishes key concepts related to stress, monitoring of one's mood, and ways in which one's mood influences one's internal thoughts and external environment; three 3-session modules correspond with key cognitive-behavioral elements: pleasant activities, thoughts, and social support/contact with others; a 1-session summary reviews content and identifies areas for future use of MB skills. Throughout MB, mood management skills are integrated using psycho-educational activities that encourage participants to understand connections between their mood and their activities, thoughts, and contacts with others.
  Arms: MB 1-on-1 Only
Behavioral: Mothers and Babies Plus Text — MB 1-on-1 along with text enhancements, both in English and Spanish. These texts focus on: a) skill reinforcement (e.g., Some thoughts just come to us, but we can make a conscious effort to think of positive thoughts.); b) homework reminders (e.g., What pleasant activity will you try today?), and c) self-monitoring (e.g., On a scale of 1-9, how would you rate your mood?). These texts will be linked with the 12 MB sessions. Specifically, after completing each in-person session, 3 texts will be sent by a home visitor to her client; one text will focus on skill reinforcement, one will be a homework reminder, and one will focus on self-monitoring.
  Arms: MB 1-on-1 Plus TEXT

SUMMARY:
This project is aimed at enhancing the effectiveness and scalability of the Mothers and Babies 1-on-1 Course (MB) among home visiting programs. MB is a manualized 12-session postpartum depression prevention intervention guided by cognitive-behavioral therapy and attachment theory. Each session lasts 15-20 minutes and is delivered as part of a regularly scheduled home visit. Previous MB trials suggest that the intervention is less successful for women who exhibit smaller changes in hypothesized intervention mechanisms and less fully engaged in completion of personal projects. This study will determine the feasibility and acceptability of conducting MB-TXT, in which home visiting clients receive MB supplemented by a series of weekly text messages focused on skill reinforcement, personal project reminders, and self-monitoring of depressive symptoms. The investigators will also calculate a preliminary effect size that could be used to calculate sample size necessary for a future fully powered randomized controlled trial that examines MB-TXT efficacy. The investigators will use a stepped wedge design-a form of randomized controlled trial that involves sequential, but random, roll-out of the intervention over multiple time periods. The investigators have created two HV program clusters. Both clusters will initially implement MB 1-on-1 and will recruit MB participants for one quarter (i.e., three months) before crossing over to recruit MB-TXT participants for one quarter. MB-TXT's core curriculum is identical to MB 1-on-1 and adds a series of text messages throughout the curriculum. Feasibility and acceptability data will be collected from clients and home visitors to assess percentages of received text messages, home visitor adherence to sending texts at specified intervals, and clients' perceptions of text message utility and clarity. If the investigators are able to integrate MB-TXT and home visiting programs and generate improved mental health outcomes for clients, the investigators will be prepared to replicate this intervention across home visiting programs nationally at a time when home visiting as a service delivery model is rapidly proliferating via federal Maternal Infant and and Early Childhood Home Visiting (MIECHV) program funding.

DETAILED DESCRIPTION:
Despite the well-established negative effects of postpartum depression on mother and child, most efforts have been directed at treating women already exhibiting depressive episodes rather than prevention. Emphasis on treatment neglects the large number of women with mild to moderate depressive symptoms, in high psychosocial risk contexts, who are at risk for developing postpartum depression. Interventions exist that are efficacious in preventing the onset and worsening of depression among perinatal women. In particular, the PI and colleagues have demonstrated that the Mothers and Babies Course (MB) prevents the worsening of depressive symptoms and onset of new major depressive episodes.

Prior MB trials suggest the intervention is less successful for women who exhibit smaller changes in hypothesized intervention mechanisms and less fully engage in homework completion between sessions-a core component of cognitive-behavioral therapy (CBT) interventions like MB. Previous postpartum depression preventive interventions-including MB-have neglected to intervene with partners of pregnant women, despite the growing recognition that paternal depression also exerts influence on children's social-emotional development and occurs in a similar time-frame. Thus, in an otherwise successful intervention, these limitations-mixed success in improving hypothesized intervention mechanisms and limited engagement of fathers-may mitigate intervention efficacy. The investigators hypothesize that core MB modules will prevent onset of major depressive episodes and worsening of depressive symptoms. The investigators also conceptualize that relationships between MB modules and maternal mental health outcomes will be mediated by mechanisms that are the direct focus of MB content.

This study addresses these limitations. The investigators will collaborate with 10-12 home visiting (HV) programs serving primarily low-income women. HV is an ideal setting for this study given the large numbers of perinatal women they serve and will build on existing relationships with HV programs in Illinois. In Phase 1, the investigators will recruit 108 pregnant women for a randomized controlled trial (RCT) in which half the participants will receive MB and half will receive MB with a text message enhancement (MB-TXT). MB-TXT will provide reinforcement of key MB skills that are linked to hypothesized mechanisms of change, promote completion of MB personal projects (homework), and facilitate self-monitoring of one's mood.

Aim 1. To determine the feasibility and acceptability of conducting the MB-TXT intervention protocol across three HV programs in preparation for a larger fully powered RCT. Using MB text messages already developed by Co-I Barrera, we will collect data on home visitor adherence to delivering text messages at specified intervals, percentage of clients responding to text messages, and client comprehension of text messages as well as perceptions of text messages' utility.

Aim 2. To calculate a preliminary effect size that could be used, along with other relevant data, to calculate sample size for a future fully powered RCT.

H1. Women receiving MB-TXT will exhibit greater reductions in depressive symptoms, compared to women receiving MB.

H2. Women receiving MB-TXT will experience greater changes in hypothesized intervention mechanisms compared to women receiving MB-specifically, fewer negative cognitions and increased behavioral activation, use of social support networks, and mood regulation.

H3. Women who participate in MB-TXT will report greater completion of personal projects.

ELIGIBILITY:
Inclusion Criteria:

English or Spanish-speaking women >16 years old enrolled in participating home visiting programs who are in their 1st or 2nd or 3rd Trimester will be eligible for enrollment

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2017-06-07 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Text messages read by HV clients | Post Intervention at 6 months
  Measured by calculating the percentage of text messages responded to by clients.
Home Visitor Adherence to MB-TXT protocol | Post Intervention at 6 months
  will be measured by using the archived data from HealthySMS to calculate the percentage of texts sent at the appropriate intervals
Client completion of personal projects | Post Intervention at 6 months
  will be measured by asking home visitors to respond to a REDCap survey item after completing each MB session to assess if clients came to the session having completed their personal project.
Client perceived utility and comprehension of text messages | Post Intervention at 6 months
  will be measured by asking home visitors to rate the extent to which each of the 3 text messages received between sessions was a) useful and b) easy to understand. Questions will be on a 4-point Likert Scale and will be asked of clients at the end of each MB session.

SECONDARY OUTCOMES:
Depressive Symptoms | Baseline and Post Intervention at 6 and 9 months
  will be assessed using the Beck Depression Inventory-II (BDI),100 a 21-item self-report measure of depressive symptoms to assess severity of depressive symptoms consistent with Diagnostic and Statistical Manual (DSM)-IV symptom criteria. The BDI has excellent internal reliability for outpatient samples and its construct validity has been established.
Cognitive Structuring | Baseline and Post Intervention at 6 and 9 months
  will be measures using the Experiences Questionnaire a 20-item self-report scale measuring decentering and rumination, which has demonstrated strong internal consistency in studies examining effects of interventions that incorporate cognitive restructuring.
Behavioral Activation | Baseline and Post Intervention at 6 and 9 months
  will be measured using the Behavioral Activation Depression Scale, a 25-item, four subscale self-report with strong psychometric properties. The four subscales assess activation, avoidance/rumination, work/school impairment, and social impairment. We will also use a brief checklist adapted from the Pleasant Events Schedule, a psychometrically strong questionnaire. This 25 item self-report contains a list of pleasant events relevant to low-income pregnant women and assesses the extent to which subject's engaged in, and experienced pleasure from, these activities.
Social Support | Baseline and Post Intervention at 6 and 9 months
  19-item Medical Outcomes Study Social Support Survey. This self-administered survey includes an overall functional social support index, as well as four functional support subscales: affectionate, emotional/informational, tangible, and positive social interaction.
Mood regulation | Baseline and Post Intervention at 6 and 9 months
  will be measured using the Negative Mood Regulation Scale (NMRS).The NMRS assesses an individual's expectancy that some behavior or cognition will alleviate a negative mood state. For each question, respondents use a five-point scale from "very much disagree" to "very much agree" to indicate what they believe they can do when they are disappointed or experiencing a negative mood. The scale has demonstrated excellent internal consistency, good test-retest reliability, and correlational evidence of both convergent and discriminant validity with constructs such as depressive symptoms and locus of control, respectively.
Mothers and Babies Skill Utilization | Baseline and Post Intervention at 6 and 9 months
  will be assessed using items developed the study investigators to assess participants utilization of the skills learned in the 12 MB sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Darius Tandon, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Evans J, Heron J, Francomb H, Oke S, Golding J. Cohort study of depressed mood during pregnancy and after childbirth. BMJ. 2001 Aug 4;323(7307):257-60. doi: 10.1136/bmj.323.7307.257. PMID 11485953
- [Background] Gaynes BN, Gavin N, Meltzer-Brody S, Lohr KN, Swinson T, Gartlehner G, Brody S, Miller WC. Perinatal depression: prevalence, screening accuracy, and screening outcomes. Evid Rep Technol Assess (Summ). 2005 Feb;(119):1-8. doi: 10.1037/e439372005-001. No abstract available. PMID 15760246
- [Background] Moses-Kolko EL, Roth EK. Antepartum and postpartum depression: healthy mom, healthy baby. J Am Med Womens Assoc (1972). 2004 Summer;59(3):181-91. PMID 15354371
- [Background] Segre LS, O'Hara MW, Arndt S, Stuart S. The prevalence of postpartum depression: the relative significance of three social status indices. Soc Psychiatry Psychiatr Epidemiol. 2007 Apr;42(4):316-21. doi: 10.1007/s00127-007-0168-1. Epub 2007 Feb 13. PMID 17370048
- [Background] Robertson E, Grace S, Wallington T, Stewart DE. Antenatal risk factors for postpartum depression: a synthesis of recent literature. Gen Hosp Psychiatry. 2004 Jul-Aug;26(4):289-95. doi: 10.1016/j.genhosppsych.2004.02.006. PMID 15234824
- [Background] Beebe B, Jaffe J, Buck K, Chen H, Cohen P, Blatt S, Kaminer T, Feldstein S, Andrews H. Six-week postpartum maternal self-criticism and dependency and 4-month mother-infant self- and interactive contingencies. Dev Psychol. 2007 Nov;43(6):1360-76. doi: 10.1037/0012-1649.43.6.1360. PMID 18020817
- [Background] Murray L, Cooper PJ, Wilson A, Romaniuk H. Controlled trial of the short- and long-term effect of psychological treatment of post-partum depression: 2. Impact on the mother-child relationship and child outcome. Br J Psychiatry. 2003 May;182:420-7. PMID 12724245
- [Background] National Research Council (US) and Institute of Medicine (US) Committee on the Prevention of Mental Disorders and Substance Abuse Among Children, Youth, and Young Adults: Research Advances and Promising Interventions; O'Connell ME, Boat T, Warner KE, editors. Preventing Mental, Emotional, and Behavioral Disorders Among Young People: Progress and Possibilities. Washington (DC): National Academies Press (US); 2009. Available from http://www.ncbi.nlm.nih.gov/books/NBK32775/ PMID 20662125
- [Background] Dave S, Sherr L, Senior R, Nazareth I. Associations between paternal depression and behaviour problems in children of 4-6 years. Eur Child Adolesc Psychiatry. 2008 Aug;17(5):306-15. doi: 10.1007/s00787-007-0672-6. Epub 2008 Mar 25. PMID 18365134
- [Background] Ramchandani PG, Stein A, O'Connor TG, Heron J, Murray L, Evans J. Depression in men in the postnatal period and later child psychopathology: a population cohort study. J Am Acad Child Adolesc Psychiatry. 2008 Apr;47(4):390-398. doi: 10.1097/CHI.0b013e31816429c2. PMID 18388761
- [Background] Fletcher RJ, Feeman E, Garfield C, Vimpani G. The effects of early paternal depression on children's development. Med J Aust. 2011 Dec 19;195(11-12):685-9. doi: 10.5694/mja11.10192. PMID 22171866
- [Background] Davis RN, Davis MM, Freed GL, Clark SJ. Fathers' depression related to positive and negative parenting behaviors with 1-year-old children. Pediatrics. 2011 Apr;127(4):612-8. doi: 10.1542/peds.2010-1779. Epub 2011 Mar 14. PMID 21402627
- [Background] Tandon SD, Perry DF, Mendelson T, Kemp K, Leis JA. Preventing perinatal depression in low-income home visiting clients: a randomized controlled trial. J Consult Clin Psychol. 2011 Oct;79(5):707-12. doi: 10.1037/a0024895. PMID 21806298
- [Background] Tandon SD, Leis JA, Mendelson T, Perry DF, Kemp K. Six-month outcomes from a randomized controlled trial to prevent perinatal depression in low-income home visiting clients. Matern Child Health J. 2014 May;18(4):873-81. doi: 10.1007/s10995-013-1313-y. PMID 23793487
- [Background] Mendelson T, Leis JA, Perry DF, Stuart EA, Tandon SD. Impact of a preventive intervention for perinatal depression on mood regulation, social support, and coping. Arch Womens Ment Health. 2013 Jun;16(3):211-8. doi: 10.1007/s00737-013-0332-4. Epub 2013 Mar 2. PMID 23456540
- [Background] Muñoz RF, Le H-N, Ippen CG, et al. Prevention of postpartum depression in low-income women: Development of the Mamás y Bebés/Mothers and Babies course. Cognitive and Behavioral Practice. 2007;14(1):70-83
- [Background] Le HN, Perry DF, Stuart EA. Randomized controlled trial of a preventive intervention for perinatal depression in high-risk Latinas. J Consult Clin Psychol. 2011 Apr;79(2):135-41. doi: 10.1037/a0022492. PMID 21319897
- [Background] Gutierrez-Galve L, Stein A, Hanington L, Heron J, Ramchandani P. Paternal depression in the postnatal period and child development: mediators and moderators. Pediatrics. 2015 Feb;135(2):e339-47. doi: 10.1542/peds.2014-2411. Epub 2015 Jan 5. PMID 25560437
- [Background] Garfield CF, Duncan G, Rutsohn J, McDade TW, Adam EK, Coley RL, Chase-Lansdale PL. A longitudinal study of paternal mental health during transition to fatherhood as young adults. Pediatrics. 2014 May;133(5):836-43. doi: 10.1542/peds.2013-3262. Epub 2014 Apr 14. PMID 24733877
- [Background] American Psychiatric Association. Diagnostic and Statistical Manual of Mental Disorders:: DSM-5. ManMag; 2003
- [Background] Howell EA, Mora PA, Horowitz CR, Leventhal H. Racial and ethnic differences in factors associated with early postpartum depressive symptoms. Obstet Gynecol. 2005 Jun;105(6):1442-50. doi: 10.1097/01.AOG.0000164050.34126.37. PMID 15932842
- [Background] Mora PA, Bennett IM, Elo IT, Mathew L, Coyne JC, Culhane JF. Distinct trajectories of perinatal depressive symptomatology: evidence from growth mixture modeling. Am J Epidemiol. 2009 Jan 1;169(1):24-32. doi: 10.1093/aje/kwn283. Epub 2008 Nov 10. PMID 19001135
- [Background] Bennett HA, Einarson A, Taddio A, Koren G, Einarson TR. Prevalence of depression during pregnancy: systematic review. Obstet Gynecol. 2004 Apr;103(4):698-709. doi: 10.1097/01.AOG.0000116689.75396.5f. PMID 15051562
- [Background] Dolbier CL, Rush TE, Sahadeo LS, Shaffer ML, Thorp J; Community Child Health Network Investigators. Relationships of race and socioeconomic status to postpartum depressive symptoms in rural African American and non-Hispanic white women. Matern Child Health J. 2013 Sep;17(7):1277-87. doi: 10.1007/s10995-012-1123-7. PMID 22961387
- [Background] Holzman C, Eyster J, Tiedje LB, Roman LA, Seagull E, Rahbar MH. A life course perspective on depressive symptoms in mid-pregnancy. Matern Child Health J. 2006 Mar;10(2):127-38. doi: 10.1007/s10995-005-0044-0. Epub 2006 Jan 7. PMID 16400535
- [Background] Giallo R, Cooklin A, Nicholson JM. Risk factors associated with trajectories of mothers' depressive symptoms across the early parenting period: an Australian population-based longitudinal study. Arch Womens Ment Health. 2014 Apr;17(2):115-25. doi: 10.1007/s00737-014-0411-1. Epub 2014 Jan 15. PMID 24424796
- [Background] Verreault N, Da Costa D, Marchand A, Ireland K, Dritsa M, Khalife S. Rates and risk factors associated with depressive symptoms during pregnancy and with postpartum onset. J Psychosom Obstet Gynaecol. 2014 Sep;35(3):84-91. doi: 10.3109/0167482X.2014.947953. PMID 25123985
- [Background] Campbell SB, Cohn JF, Flanagan C, Popper S, Meyers T. Course and correlates of postpartum depression during the transition to parenthood. Development and psychopathology. 1992;4(01):29-47
- [Background] O'Hara M. Postpartum depression: identification and measurement in a cross-cultural context. Perinatal psychiatry: Use and misuse of the Edinburgh Postnatal Depression Scale. London: Gaskell. 1994:145-168.
- [Background] Weinberg MK, Tronick EZ, Beeghly M, Olson KL, Kernan H, Riley JM. Subsyndromal depressive symptoms and major depression in postpartum women. Am J Orthopsychiatry. 2001 Jan;71(1):87-97. doi: 10.1037/0002-9432.71.1.87. PMID 11271721
- [Background] Wisner KL, Perel JM, Peindl KS, Hanusa BH. Timing of depression recurrence in the first year after birth. J Affect Disord. 2004 Mar;78(3):249-52. doi: 10.1016/S0165-0327(02)00305-1. PMID 15013250
- [Background] Lindahl V, Pearson JL, Colpe L. Prevalence of suicidality during pregnancy and the postpartum. Arch Womens Ment Health. 2005 Jun;8(2):77-87. doi: 10.1007/s00737-005-0080-1. Epub 2005 May 11. PMID 15883651
- [Background] Logsdon MC, Wisner K, Sit D, Luther JF, Wisniewski SR. Depression treatment and maternal functioning. Depress Anxiety. 2011 Nov;28(11):1020-6. doi: 10.1002/da.20892. Epub 2011 Sep 2. PMID 21898714
- [Background] O'Hara MW. Postpartum depression: what we know. J Clin Psychol. 2009 Dec;65(12):1258-69. doi: 10.1002/jclp.20644. PMID 19827112
- [Background] Lovejoy MC, Graczyk PA, O'Hare E, Neuman G. Maternal depression and parenting behavior: a meta-analytic review. Clin Psychol Rev. 2000 Aug;20(5):561-92. doi: 10.1016/s0272-7358(98)00100-7. PMID 10860167
- [Background] Foster CJ, Garber J, Durlak JA. Current and past maternal depression, maternal interaction behaviors, and children's externalizing and internalizing symptoms. J Abnorm Child Psychol. 2008 May;36(4):527-37. doi: 10.1007/s10802-007-9197-1. Epub 2007 Dec 11. PMID 18071896
- [Background] Chronicity of maternal depressive symptoms, maternal sensitivity, and child functioning at 36 months. NICHD Early Child Care Research Network. Dev Psychol. 1999 Sep;35(5):1297-310. doi: 10.1037//0012-1649.35.5.1297. PMID 10493655
- [Background] Horwitz SM, Briggs-Gowan MJ, Storfer-Isser A, Carter AS. Prevalence, correlates, and persistence of maternal depression. J Womens Health (Larchmt). 2007 Jun;16(5):678-91. doi: 10.1089/jwh.2006.0185. PMID 17627403
- [Background] Siu AL; US Preventive Services Task Force (USPSTF); Bibbins-Domingo K, Grossman DC, Baumann LC, Davidson KW, Ebell M, Garcia FA, Gillman M, Herzstein J, Kemper AR, Krist AH, Kurth AE, Owens DK, Phillips WR, Phipps MG, Pignone MP. Screening for Depression in Adults: US Preventive Services Task Force Recommendation Statement. JAMA. 2016 Jan 26;315(4):380-7. doi: 10.1001/jama.2015.18392. PMID 26813211
- [Background] Vázquez FL, Muñoz RF, Blanco V, López M. Validation of Muñoz's Mood Screener in a nonclinical Spanish population. European Journal of Psychological Assessment. 2008;24(1):57-64.
- [Background] Bennett IM, Marcus SC, Palmer SC, Coyne JC. Pregnancy-related discontinuation of antidepressants and depression care visits among Medicaid recipients. Psychiatr Serv. 2010 Apr;61(4):386-91. doi: 10.1176/ps.2010.61.4.386. PMID 20360278
- [Background] Abrams LS, Dornig K, Curran L. Barriers to service use for postpartum depression symptoms among low-income ethnic minority mothers in the United States. Qual Health Res. 2009 Apr;19(4):535-51. doi: 10.1177/1049732309332794. PMID 19299758
- [Background] Dennis CL, Chung-Lee L. Postpartum depression help-seeking barriers and maternal treatment preferences: a qualitative systematic review. Birth. 2006 Dec;33(4):323-31. doi: 10.1111/j.1523-536X.2006.00130.x. PMID 17150072
- [Background] O'Mahen HA, Flynn HA. Preferences and perceived barriers to treatment for depression during the perinatal period. J Womens Health (Larchmt). 2008 Oct;17(8):1301-9. doi: 10.1089/jwh.2007.0631. PMID 18816202
- [Background] Kim JJ, La Porte LM, Corcoran M, Magasi S, Batza J, Silver RK. Barriers to mental health treatment among obstetric patients at risk for depression. Am J Obstet Gynecol. 2010 Mar;202(3):312.e1-5. doi: 10.1016/j.ajog.2010.01.004. PMID 20207252
- [Background] Smith MV, Shao L, Howell H, Wang H, Poschman K, Yonkers KA. Success of mental health referral among pregnant and postpartum women with psychiatric distress. Gen Hosp Psychiatry. 2009 Mar-Apr;31(2):155-62. doi: 10.1016/j.genhosppsych.2008.10.002. Epub 2008 Dec 3. PMID 19269536
- [Background] U.S. Department of Health and Human Services, Maternal and Child Health Bureau. Women's Health USA 2013. http://mchb.hrsa.gov/whusa13/health-services-utilization/pdf/mhcu.pdf. Accessed October 1.
- [Background] Mayberry LJ, Horowitz JA, Declercq E. Depression symptom prevalence and demographic risk factors among U.S. women during the first 2 years postpartum. J Obstet Gynecol Neonatal Nurs. 2007 Nov-Dec;36(6):542-9. doi: 10.1111/j.1552-6909.2007.00191.x. PMID 17973697
- [Background] Cuijpers P, de Graaf R, van Dorsselaer S. Minor depression: risk profiles, functional disability, health care use and risk of developing major depression. J Affect Disord. 2004 Apr;79(1-3):71-9. doi: 10.1016/S0165-0327(02)00348-8. PMID 15023482
- [Background] Wagner HR, Burns BJ, Broadhead WE, Yarnall KS, Sigmon A, Gaynes BN. Minor depression in family practice: functional morbidity, co-morbidity, service utilization and outcomes. Psychol Med. 2000 Nov;30(6):1377-90. doi: 10.1017/s0033291799002998. PMID 11097078
- [Background] Dennis CL, Dowswell T. Psychosocial and psychological interventions for preventing postpartum depression. Cochrane Database Syst Rev. 2013 Feb 28;2013(2):CD001134. doi: 10.1002/14651858.CD001134.pub3. PMID 23450532
- [Background] Lewinsohn P, Muñoz R, Youngren M, Zeiss A. Control Your Depression. Reducing Depression through Learning Self-Control Techniques, Relaxation Training, Pleasant Activities, Social Skills, Constructed Thinking, Planning Ahead and More. New York: Simon & Schuster Inc; 1986
- [Background] Ainsworth M, Blehar M, Waters E. Wall. s.(1978). Patterns of attachment: A psychological study of the strange situation
- [Background] Bowlby J. Attachment and loss. Vol 3: Basic books; 1980
- [Background] McFarlane E, Burrell L, Duggan A, Tandon D. Outcomes of a Randomized Trial of a Cognitive Behavioral Enhancement to Address Maternal Distress in Home Visited Mothers. Matern Child Health J. 2017 Mar;21(3):475-484. doi: 10.1007/s10995-016-2125-7. PMID 27535131
- [Background] Madden M. Technology use by different income groups. 2013; http://www.pewinternet.org/2013/05/29/technology-use-by-different-income-groups/. Accessed February 2, 2016.
- [Background] Anderson M. Technology device ownership: 2015. 2015; http://www.pewinternet.org/2015/10/29/technology-device-ownership-2015/. Accessed February 2, 2016.
- [Background] Fjeldsoe BS, Marshall AL, Miller YD. Behavior change interventions delivered by mobile telephone short-message service. Am J Prev Med. 2009 Feb;36(2):165-73. doi: 10.1016/j.amepre.2008.09.040. PMID 19135907
- [Background] Kannisto KA, Koivunen MH, Valimaki MA. Use of mobile phone text message reminders in health care services: a narrative literature review. J Med Internet Res. 2014 Oct 17;16(10):e222. doi: 10.2196/jmir.3442. PMID 25326646
- [Background] Broom MA, Ladley AS, Rhyne EA, Halloran DR. Feasibility and Perception of Using Text Messages as an Adjunct Therapy for Low-Income, Minority Mothers With Postpartum Depression. JMIR Ment Health. 2015 Mar 16;2(1):e4. doi: 10.2196/mental.4074. eCollection 2015 Jan-Mar. PMID 26543910
- [Background] Soltani H, Furness PJ, Arden MA, McSeveny K, Garland C, Sustar H, Dearden A. Women's and Midwives' Perspectives on the Design of a Text Messaging Support for Maternal Obesity Services: An Exploratory Study. J Obes. 2012;2012:835464. doi: 10.1155/2012/835464. Epub 2012 Jul 26. PMID 22900153
- [Background] Cormick G, Kim NA, Rodgers A, Gibbons L, Buekens PM, Belizan JM, Althabe F. Interest of pregnant women in the use of SMS (short message service) text messages for the improvement of perinatal and postnatal care. Reprod Health. 2012 Aug 6;9:9. doi: 10.1186/1742-4755-9-9. PMID 22866753
- [Background] Waring ME, Moore Simas TA, Xiao RS, Lombardini LM, Allison JJ, Rosal MC, Pagoto SL. Pregnant women's interest in a website or mobile application for healthy gestational weight gain. Sex Reprod Healthc. 2014 Dec;5(4):182-4. doi: 10.1016/j.srhc.2014.05.002. Epub 2014 May 14. PMID 25433828
- [Background] Poorman E, Gazmararian J, Parker RM, Yang B, Elon L. Use of text messaging for maternal and infant health: a systematic review of the literature. Matern Child Health J. 2015 May;19(5):969-89. doi: 10.1007/s10995-014-1595-8. PMID 25081242
- [Background] Paulson JF, Bazemore SD. Prenatal and postpartum depression in fathers and its association with maternal depression: a meta-analysis. JAMA. 2010 May 19;303(19):1961-9. doi: 10.1001/jama.2010.605. PMID 20483973
- [Background] Bronte-Tinkew J, Moore KA, Matthews G, Carrano J. Symptoms of major depression in a sample of fathers of infants sociodemographic correlates and links to father involvement. Journal of family Issues. 2007;28(1):61-99.
- [Background] Paulson JF, Keefe HA, Leiferman JA. Early parental depression and child language development. J Child Psychol Psychiatry. 2009 Mar;50(3):254-62. doi: 10.1111/j.1469-7610.2008.01973.x. Epub 2008 Oct 23. PMID 19175819
- [Background] Dennis CL, Dowswell T. Interventions (other than pharmacological, psychosocial or psychological) for treating antenatal depression. Cochrane Database Syst Rev. 2013 Jul 31;2013(7):CD006795. doi: 10.1002/14651858.CD006795.pub3. PMID 23904069
- [Background] Barlow J, Smailagic N, Huband N, Roloff V, Bennett C. Group-based parent training programmes for improving parental psychosocial health. Cochrane Database Syst Rev. 2014 May 17;2014(5):CD002020. doi: 10.1002/14651858.CD002020.pub4. PMID 24838729
- [Background] Schmit S, Schott L, Pavetti L, Matthews H. Effective, Evidence-Based Home Visiting Programs in Every State at Risk if Congress Does Not Extend Funding. 2015; http://www.cbpp.org/research/effective-evidence-based-home-visiting-programs-in-every-state-at-risk-if-congress-does-not. Accessed February 10, 2016.
- [Background] Avellar S, Paulsell D, Sama-Miller E, Grosso PD, Akers L, Kleinman R. Home visiting evidence of effectiveness review: Executive summary. Mathematica Policy Research;2013
- [Background] U.S. Department of Health and Human Services, Administration for Children and Families, Office of Planning and Evaluation. Depression in the Lives of Early Head Start Families: Research to Practice Brief. 2006; http://www.acf.hhs.gov/programs/opre/resource/depression-in-the-lives-of-early-head-start-families-research-to-practice. Accessed January 15, 2014. Accessed January 15, 2016
- [Background] U.S. Department of Health and Human Services, Health Resources and Services Administration, Maternal and Child Health Bureau. A Comprehensive Approach for Community-Based Programs to Address Intimate Partner Violence and Perinatal Depression. 2013; http://mchb.hrsa.gov/pregnancyandbeyond/depression/partnerviolence/partnerviolenceandperinataldepression.pdf.Accessed February 10 2016.
- [Background] Prevent Child Abuse America. Healthy Families America Critical Elements. 2001; http://www.healthyfamiliesamerica.org/downloads/critical_elements_rationale.pdf. Accessed January 15, 2016.
- [Background] Ammerman RT, Putnam FW, Bosse NR, Teeters AR, Van Ginkel JB. Maternal Depression in Home Visitation: A Systematic Review. Aggress Violent Behav. 2010 May;15(3):191-200. doi: 10.1016/j.avb.2009.12.002. PMID 20401324
- [Background] Ammerman RT, Putnam FW, Altaye M, Chen L, Holleb LJ, Stevens J, Short JA, Van Ginkel JB. Changes in depressive symptoms in first time mothers in home visitation. Child Abuse Negl. 2009 Mar;33(3):127-38. doi: 10.1016/j.chiabu.2008.09.005. Epub 2009 Mar 27. PMID 19328548
- [Background] Chazan-Cohen R, Ayoub C, Pan BA, Roggman L, Raikes H, Mckelvey L, Whiteside-Mansell L, Hart A. It takes time: Impacts of Early Head Start that lead to reductions in maternal depression two years later. Infant Ment Health J. 2007 Mar;28(2):151-170. doi: 10.1002/imhj.20127. PMID 28640556
- [Background] Tandon SD, Parillo KM, Jenkins C, Duggan AK. Formative evaluation of home visitors' role in addressing poor mental health, domestic violence, and substance abuse among low-income pregnant and parenting women. Matern Child Health J. 2005 Sep;9(3):273-83. doi: 10.1007/s10995-005-0012-8. PMID 16240078
- [Background] Garfield CF, Lee Y, Kim HN. Paternal and maternal concerns for their very low-birth-weight infants transitioning from the NICU to home. J Perinat Neonatal Nurs. 2014 Oct-Dec;28(4):305-12. doi: 10.1097/JPN.0000000000000021. PMID 24927295
- [Background] Kim HN, Garfield C, Lee YS. Paternal and Maternal Information and Communication Technology Usage as Their Very Low Birth Weight Infants Transition Home From the NICU. International Journal of Human-Computer Interaction. 2015;31(1):44-54.
- [Background] Cox JL, Holden JM, Sagovsky R. Detection of postnatal depression. Development of the 10-item Edinburgh Postnatal Depression Scale. Br J Psychiatry. 1987 Jun;150:782-6. doi: 10.1192/bjp.150.6.782. PMID 3651732
- [Background] Meijer JL, Beijers C, van Pampus MG, Verbeek T, Stolk RP, Milgrom J, Bockting CL, Burger H. Predictive accuracy of Edinburgh postnatal depression scale assessment during pregnancy for the risk of developing postpartum depressive symptoms: a prospective cohort study. BJOG. 2014 Dec;121(13):1604-10. doi: 10.1111/1471-0528.12759. Epub 2014 Apr 7. PMID 24703235
- [Background] Rush AJ, Trivedi MH, Ibrahim HM, Carmody TJ, Arnow B, Klein DN, Markowitz JC, Ninan PT, Kornstein S, Manber R, Thase ME, Kocsis JH, Keller MB. The 16-Item Quick Inventory of Depressive Symptomatology (QIDS), clinician rating (QIDS-C), and self-report (QIDS-SR): a psychometric evaluation in patients with chronic major depression. Biol Psychiatry. 2003 Sep 1;54(5):573-83. doi: 10.1016/s0006-3223(02)01866-8. PMID 12946886
- [Background] Trivedi MH, Rush AJ, Ibrahim HM, Carmody TJ, Biggs MM, Suppes T, Crismon ML, Shores-Wilson K, Toprac MG, Dennehy EB, Witte B, Kashner TM. The Inventory of Depressive Symptomatology, Clinician Rating (IDS-C) and Self-Report (IDS-SR), and the Quick Inventory of Depressive Symptomatology, Clinician Rating (QIDS-C) and Self-Report (QIDS-SR) in public sector patients with mood disorders: a psychometric evaluation. Psychol Med. 2004 Jan;34(1):73-82. doi: 10.1017/s0033291703001107. PMID 14971628
- [Background] Fresco DM, Moore MT, van Dulmen MH, Segal ZV, Ma SH, Teasdale JD, Williams JM. Initial psychometric properties of the experiences questionnaire: validation of a self-report measure of decentering. Behav Ther. 2007 Sep;38(3):234-46. doi: 10.1016/j.beth.2006.08.003. Epub 2007 Apr 24. PMID 17697849
- [Background] Kanter JW, Mulick PS, Busch AM, Berlin KS, Martell CR. The Behavioral Activation for Depression Scale (BADS): psychometric properties and factor structure. Journal of Psychopathology and Behavioral Assessment. 2007;29(3):191-202.
- [Background] Kanter JW, Rusch LC, Busch AM, Sedivy SK. Validation of the Behavioral Activation for Depression Scale (BADS) in a community sample with elevated depressive symptoms. Journal of Psychopathology and Behavioral Assessment. 2009;31(1):36-42.
- [Background] Teri L, Lewinsohn P. Modification of the Pleasant and Unpleasant Events Schedules for use with the elderly. J Consult Clin Psychol. 1982 Jun;50(3):444-5. doi: 10.1037//0022-006x.50.3.444. No abstract available. PMID 7096747
- [Background] Sherbourne CD, Stewart AL. The MOS social support survey. Soc Sci Med. 1991;32(6):705-14. doi: 10.1016/0277-9536(91)90150-b. PMID 2035047
- [Background] Catanzaro SJ, Greenwood G. Expectancies for negative mood regulation, coping, and dysphoria among college students. Journal of Counseling Psychology. 1994;41(1):34.
- [Background] Catanzaro SJ, Mearns J. Measuring generalized expectancies for negative mood regulation: initial scale development and implications. J Pers Assess. 1990 Summer;54(3-4):546-63. doi: 10.1080/00223891.1990.9674019. PMID 2348341
- [Background] Garfield CF, Isacco III AJ. Urban fathers' involvement in their child's health and healthcare. Psychology of Men & Masculinity. 2012;13(1):32.
- [Background] Garfield CF, Isacco A. Fathers and the well-child visit. Pediatrics. 2006 Apr;117(4):e637-45. doi: 10.1542/peds.2005-1612. PMID 16585280
- [Background] Tandon SD, Parillo KM, Keefer M. Hispanic women's perceptions of patient-centeredness during prenatal care: a mixed-method study. Birth. 2005 Dec;32(4):312-7. doi: 10.1111/j.0730-7659.2005.00389.x. PMID 16336373
- [Background] Tandon SD, Mercer CD, Saylor EL, Duggan AK. Paraprofessional home visitors' perspectives on addressing poor mental health, substance abuse, and domestic violence: A qualitative study. Early Childhood Research Quarterly. 2008;23(3):419-428
- [Background] Mance GA, Mendelson T, Byrd B, Jones J, Tandon D. Utilizing community-based participatory research to adapt a mental health intervention for African American emerging adults. Prog Community Health Partnersh. 2010 Summer;4(2):131-40. doi: 10.1353/cpr.0.0112. PMID 20543488
- [Background] Crane DR, Middleton KC, Bean RA. Establishing criterion scores for the Kansas marital satisfaction scale and the revised dyadic adjustment scale. American Journal of Family Therapy. 2000;28(1):53-60.
- [Background] Snow K, Thalji L, Derecho A, et al. Early Childhood Longitudinal Study, Birth Cohort (ECLS-B), Preschool Year Data File User's Manual (2005-06)(NCES 2008-024). Washington, DC: National Center for Education Statistics, Institute of Education Sciences, US Department of Education. 2007:1-190.
- [Background] Procidano ME, Heller K. Measures of perceived social support from friends and from family: three validation studies. Am J Community Psychol. 1983 Feb;11(1):1-24. doi: 10.1007/BF00898416. PMID 6837532
- [Derived] Barrera AZ, Hamil J, Tandon D. Integrating SMS Text Messages Into a Preventive Intervention for Postpartum Depression Delivered via In-Home Visitation Programs: Feasibility and Acceptability Study. JMIR Form Res. 2021 Nov 18;5(11):e30995. doi: 10.2196/30995. PMID 34792478